CLINICAL TRIAL: NCT03562962
Title: Assessing the Mechanism of Change of Functional Analytic Psychotherapy: An Analysis of a Process-Driven Behavioral Intervention
Brief Title: Assessing the Mechanism of Change of Functional Analytic Psychotherapy
Acronym: FAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Reno (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1116749-3
Record Dates: First submitted 2018-03-27; First posted 2018-06-20 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-06

CONDITIONS: Interpersonal Functioning; Psychological Distress
Keywords: Functional Analytic Psychotherapy; Process-Outcome Psychotherapies; Mechanism of change; Interpersonal Functioning; Psychological Distress; Contingencies of reinforcement

STUDY DESIGN:
Intervention Model Description: A concurrent experimental multiple baseline design (MBL) across participants with a follow-up phase will be conducted (A/B/Follow-up). Concurrent MBL controls historical factors and other threats to internal validity by sequentially introducing the treatment phase. The latter requires that the length of the baselines varies between participants. Additionally, the MBL allows comparing behavioral data among individuals across different or similar conditions, showing whether extraneous variables affect the participants in the same manner or not. The between-series comparisons control for threats to external and internal validity that might affect individuals in the same study.
Masking Description: An independent blind Research Assistant (RA) will score and record the data from questionnaires administered before and after therapeutic sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Functional Analytic Psychotherapy (Other): Within the baseline (A), Supportive Listening (SL) will be provided, which has been widely utilized in randomized control trials (Cuijpers et al., 2012), including the only Randomized Control Trial (RCT) conducted in FAP (Maitland & Gaynor, 2016), as a control condition. SL is defined as "a psychological treatment in which therapists do not engage in any therapeutic strategies other than active listening and offering support, focusing on participants' problems and concerns" (Cuijpers et al., 2012, p. 281). In this therapy, the therapist reflects on clients' experiences and encourage them to share emotional experiences. Therapists are prohibited from giving advice, making interpretations, and providing feedback to clients (Cuijpers et al., 2012).
  FAP will be introduced at phase B, where contingent reinforcement will be administered for increasing clients' alternative behaviors (CRB2) and differential reinforcement will be utilized to reduce clients' problem behaviors (CRB1).
  Interventions: Behavioral: Functional Analytic Psychotherapy

INTERVENTIONS:
Behavioral: Functional Analytic Psychotherapy — FAP is a therapeutic procedure based on behavior analytic principles. This approach seeks to implement procedures to manipulate the contingencies of reinforcement involved in clients' problem and alternative behaviors within the context of a meaningful therapeutic relationship that is functionally equivalent to other interpersonal contexts outside (Follette, Naugle & Linnerooth, 2000; Kohlenberg & Tsai, 1991). FAP therapists modify CRBs by implementing contingent responding (TCRB) within the therapeutic setting. That is, FAP aims to administer differential reinforcement (TCRB1) to reduce CRB1s and to provide positive reinforcement to enhance CRB2s. Based on the changes within the therapeutic setting, clients are prompted to discriminate contexts where those repertoires are likely reinforced and to generalize those responses to such environments (Kohlenberg & Tsai, 1991).
  Other Names: FAP

SUMMARY:
This study seeks to assess the mechanisms of change of Functional Analytic Psychotherapy (FAP). FAP is a process-outcome psychotherapy that focuses on the therapeutic relationship, providing services to participants presenting with difficulties in their social interactions and relationships. A multiple baseline design between four participants who report interpersonal relating difficulties and psychological distress will be conducted. Therapists will provide contingent reinforcement to clients' behavior in session with the aim of:

1. Examining the mechanisms of change of FAP via contingent responding to participants' interpersonal difficulties.
2. Determining the effectiveness of FAP on the interpersonal functioning of verbally able adults.
3. Establishing the relationship between the amount of contingent reinforcement and the changes in clients' interpersonal repertoires (proportion).

Four hypotheses will be explored in this study: (1) contingent reinforcement functions as the mechanism of change in FAP, (2) FAP implementation decreases the frequency of interpersonal problems in and out of session, (3) FAP implementation increases the frequency of interpersonal functioning in and out of session, and (4) a higher proportion of reinforcement delivered by therapist enhances clients' alternative behaviors.

DETAILED DESCRIPTION:
The interest for supporting process-outcome psychotherapies has increased in recent years. With the aim of finding parsimonious and precise interventions for specific populations under particular circumstances, clinical researchers have supported the development of principle-driven research. Studies discussed the importance of conducting translational research to identify psychotherapy mechanisms of change in order to match those interventions with psychological problems maintained by similar variables. In the long term, it is expected that process-outcome psychotherapies will reduce the burden produced by the overload of psychological interventions that share similar mechanisms of change but have been treated as independent therapeutic packages. Likewise, it is anticipated that process-outcome psychotherapies will reduce relapse frequency by targeting specific mechanisms of change. They would also enhance efficiency since they will reduce the use of therapeutic procedures that do not target the most important variables in producing therapeutic change.

Functional Analytic Psychotherapy (FAP) is a process-outcome psychotherapy that produces changes in interpersonal relating behaviors by modifying the contingencies of reinforcement of clients' behavior. Reinforcement, as a behavioral mechanism of change, explains the increment on the probability of occurrence of the behavior and its maintenance. FAP focuses on improving the effectiveness of clients' interpersonal behaviors by providing social contingencies of reinforcement to clients' responses within the therapeutic setting. Though there are several studies and reports that support the effectiveness of FAP, few studies have explored the specific mechanisms of change. Some studies have explored the effects of therapists' contingent responding to clients' ineffective behavior. However, they have lacked analyses of conditional relationships between clients and therapists' responses. This research, therefore, will provide information about the mechanism of change underlying FAP by studying the conditional relations of contingencies of reinforcement and clients' behaviors in the context of a meaningful therapeutic relationship.

Method

Study aims:

1. To examine the mechanisms of change of Functional Analytic Psychotherapy (FAP) via contingent responding to participants' interpersonal difficulties
2. To determine the effectiveness of FAP on the interpersonal functioning of verbally able adults.
3. To establish the relation between the amount of contingent reinforcement and the changes in clients' interpersonal repertoires.

Variables:

Dependent. Interpersonal relating difficulties comprise behaviors that interfere with social functioning. In Callaghan's words, "[t]hese problems are based on the function of behaviors as they impact the client's ability to form effective interpersonal relationships". Lastly, interpersonal difficulties are defined based on the effects these produce on the individual's the social environment (function). Behavior analysis identifies two types of operant functions that characterize classes of behavior: positive reinforcement, a process by which behaviors are strengthened following the delivery of a consequence, and negative reinforcement, where behaviors are strengthened by the withdrawal of a potentially aversive consequence.

Callaghan developed the Functional Idiographic Assessment Template (FIAT), a functional based classification for interpersonal difficulties. The FIAT described repertoires based on the antecedent stimulus control and the behavioral patterns (which include the contingency of reinforcement). Five functional interpersonal classes will be object of intervention in this study: (a) assertion of needs (including social support), (b) bidirectional communication, (c) conflict, (d) disclosure and interpersonal closeness (disclosing and seeking intimacy), and (e) emotional experience and expression. Problems in the FIAT classes (CRB1s) will be modified by altering the contingencies of reinforcement as specified in the description of the independent variable, aiming increasing improvements in these functional classes (CRB2s).

Independent. FAP is a therapeutic procedure based on behavior analytic principles. This approach seeks to implement procedures to manipulate the contingencies of reinforcement involved in problem and alternative behaviors within the context of a meaningful therapeutic relationship in the clinical setting that is functionally equivalent to those out-of-session.

According to the behavior analytic perspective, there are two main processes (functions of behavior) that are targeted to influence individuals' behavior: contingencies of reinforcement (process that maintains elevations or increases behavior probability) and antecedent stimulus control, which involves a set of conditions under which the responses are more likely reinforced. A discriminative stimulus (SD) indicates that reinforcement is available, whereas a Delta stimulus (SΔ) signals an extremely low probability for reinforcement of behavior. These functional relations are identified using a functional behavioral assessment. FAP intends to modify CRBs by utilizing therapists contingent responding (TCRB). That is, FAP proposed to implement differential reinforcement (TCRB1) to reduce CRB1s and to provide positive reinforcement to enhance CRB2s. Based on the changes within the therapeutic setting, clients are prompted to discriminate contexts where those repertoires are likely reinforced and generalize those responses to such environments.

Design:

A non-concurrent experimental multiple baseline design (MBL) across participants with a follow-up phase will be conducted (A/B/Follow-up). Concurrent MBL controls historical factors and other threats to internal validity by sequentially introducing the treatment phase. The latter requires that the length of the baselines varies between participants. In this study, the baselines per each participant will be assigned in this order: three sessions to the participant 1, five sessions to the participant, six sessions to participant 3, and seven sessions to participant 4.

Additionally, the MBL allows comparing behavioral data between individuals across different or similar conditions, showing whether extraneous variables affect the participants in the same manner or not. The between-series comparisons control for historical factors or other threats to external and internal validity that might affect individuals in the same study.

Within the baseline (A), Supportive Listening (SL) will be provided, which has been widely utilized in randomized control trials, including the only Randomized Control Trial (RCT) conducted in FAP (Maitland & Gaynor, 2016), as a control condition. SL is defined as "a psychological treatment in which therapists do not engage in any therapeutic strategies other than active listening and offering support, focusing on participants' problems and concerns". In this therapy, the therapist reflects on clients' experiences and encourage them to share emotional experiences. Therapists are prohibited from giving advice, making interpretations, and providing feedback to clients. FAP will be introduced at phase B, where contingent reinforcement will be administered for increasing clients' goal behaviors (CRB2) and differential reinforcement will be utilized to reduce clients' problem behaviors (CRB1).

Participants:

The study will include four participants. Based on the power analysis performed using the D_power macro, the study will have a power of .962 (high power). They will be recruited using flyers that will be posted on public billboards on University campus (University of Nevada, Reno). Third party (or snowball sampling) procedures will be also utilized. Participants will be recruited through the Psychological Services Center as well as the Student Counseling Center at the University of Nevada, Reno. A flyer with the study and contact instruction information will be provided to these sites with the aim that the potential participants initiate the contact with the researchers subsequently.

Up to 20 participants will be recruited and an eligibility assessment will be conducted by two doctoral students to determine participants enrollment. Potential participants who report interpersonal difficulties and psychological distress will be invited to enroll in the study. Interpersonal functioning will be assessed using the Functional Idiographic Assessment Template-Questionnaire Short Form (FIAT-Q-SF), and psychological distress will be evaluated utilizing the Depression Anxiety Stress Scales (DASS). A clinical interview will be conducted to validate participants' interpersonal and psychological functioning. Individuals who report current substance abuse disorder as defined by the DSM-5, suicidal plan or past suicidal attempts and history of psychotic or bipolar disorder will be excluded and referred to another psychological service provider.

Instruments and Materials:

1. Functional Idiographic Assessment Template-Questionnaire Short Form (FIAT-Q-SF): to identify participants interpersonal functioning outside the therapeutic setting.
2. Depression Anxiety Stress Scales (DASS): to identify participants psychological distress outside the therapeutic setting.
3. The Functional Analytic Psychotherapy-Intimacy Scale (FAP-IS): to identify participants' engagement in a meaningful therapeutic relationship that facilities the action of the mechanism of change in FAP.
4. Working Alliance Inventory-Short Revised (WAI-SF): to identify participants' engagement in a meaningful therapeutic relationship that facilities the action of the mechanism of change in FAP.
5. Functional Analytic Psychotherapy Rating Scale (FAPRS): The FAPRS is a coding system designed for assessing clinical interactions based on behavior analytic principles. This instrument will be employed to evaluate FAP's mechanism of change and therapists' adherence to FAP procedures.
6. Diary Card (Self-report record): to assess participant's interpersonal behaviors outside of session. This format includes three columns where participants describe the antecedents and consequences of their interpersonal behaviors.
7. Noldus Observer XT: this software allows coders to observe and code participants and therapists' behaviors in-session with the aim of assessing the mechanism of change in FAP.

Procedure:

During recruitment, potential participants will be invited to attend 1-hr and a half eligibility assessment session. Before conducting the eligibility assessment, informed consents will be discussed with potential participants according to APA and local IRB standards. Upon participants agree on research participation, interpersonal difficulties and psychological distress will be evaluated. Results of eligibility will be discussed at the end of this session. If a potential participant decides to decline or discontinue his/her participation or does not meet criteria for the study, referral options will be provided using a referral list of the psychological services center (PSC). Assessments will be conducted in the PSC by the therapists in this study.

Following enrollment, SL and clients' history assessment will be conducted (Baseline). At the first three weeks, phase B will be introduced to the first participant at session four and the intervention will be sequentially implemented to the other clients as described in the design section. FAP will be introduced to modify the functions that maintain the interpersonal relating difficulties (nine-weeks per each participant). Finally, a follow-up session will take place one month after completion of the intervention phase, and stability of behavior changes across time will be measured.

Data will be collected on a weekly basis. FIAT-Q-SF and DASS will be administered at the beginning of the session, to assess participants interpersonal functioning and psychological distress out-of-session. WAI-SF and FAP-IS will be administered at the end of therapy and place in a sealed box, to prevent responders' bias on the quality of therapeutic relationship. Scores from these questionaries' will be entered in an Excel sheet within an electronic server encrypted by a blind research assistant. In addition, participants and therapists' behaviors within the therapeutic session will be coded by three blind raters with the aim of assessing the mechanism of change of FAP and the effects of FAP in interpersonal functioning and psychological distress in the session. Video records will be kept safe in an electronic file encrypted storage and a password-protected computer.

For quality assurance, data will be monitored by the principal investigator weekly. The principal investigator will review participants case report forms and conduct meetings with the therapists to oversee the fidelity of research procedures. Adverse reactions will be assessed applying the knowledge the principal investigator has of clinical factors and behaviors that predict and indicate adverse psychological reactions. He also has a vast knowledge in FAP that allows him to detect negative unexpected effects from implementing this intervention. So far, FAP research has not found specific therapeutic factors that would trigger an immediate suspension of the research. If so, the principal investigator will inform local IRB and the study procedures would be re-evaluated or suspended.

Data Analysis Plan:

To examine the mechanisms of change of the FAP via contingent responding to participants' interpersonal difficulties (Aim 1), a state-based lag sequential analysis of participants and therapist behaviors within session will be conducted. The statistical significance of the conditional probabilities will be tested by computing z scores (adjusted residuals). The strength of the association between client and therapist's behavior will be examined by the Yule's Q statistic and a chi-squared test will be performed to identify a significant interdependence within the transitional matrix. In addition, a stack graph will be performed to analyze the relationship between the CRBs and the percentage of contingent reinforcement in the context of a meaningful relationship (FAP-IS).

Effectiveness of FAP on interpersonal difficulties of verbally able adults (Aim 2) will be examined by conducting descriptive statistics and visual inspection of participants' behaviors to compare trends between-subjects. Effect sizes will be determined by calculating Hedge's g correction of standardized effect sizes for singles case designs. A non-overlap analysis of all pairs (NAP) will be conducted as a complementary assessment of the effect sizes of participants' behaviors. In addition, a simulation modelling analysis (SMA) will be performed to establish the relation between FAP and changes in interpersonal difficulties. SMA is an alternative statistical technique that has an acceptable control of Type-I and Type-II errors to analyzed short streams of autocorrelated data, which are typically observed in single case designs. This statistical method simulates datasets similar in length and autocorrelation to the data at hand. Using a bootstrapping, SMA tests if the relationship between the intervention and the dependent variable remains when autocorrelation and data length are similar in thousand (~5000) of samples.

To establish the relation between the amount of contingent reinforcement and the changes in clients' interpersonal repertoires in session (Aim 3), the proportion of therapists' contingent responses (TCRBs) to CRBs will be calculated. TCRBs' proportion will be plotted and a visual analysis of behavioral trends between participants will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Interpersonal Difficulties: participants who endorse high scores in the Functional Idiographic Assessment Template-Questionnaire Short Form (Darrow et al., 2014) and report interpersonal dysfunction in a clinical interview based on the Functional Idiographic Assessment Template (Callaghan, 2001)
* Psychological Distress: participants who endorse indicators of depression, anxiety, stress, or general psychological distress based on the DASS-42 (Crawford & Henry, 2003) and report psychological distress in a clinical interview.
* Participants who Identify themselves as needing psychological services.

Exclusion Criteria:

* Current substance abuse.
* Current suicidal plan.
* Past suicidal attempts.
* History of psychotic or bipolar disorders.
* Participants who are taking psychiatric medication for less than six weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
Functional Idiographic Assessment Template-Questionnaire Short Form (FIAT-Q-SF) | Through study completion, an average of 1 year
  FIAT-Q-SF is a 32-items self-report in a 6-point liker scale (from -3 to +3) based on a functional analytic approach of interpersonal functioning. Items are contained in six interpersonal factors that have moderate and good reliability using Cronbach's alpha: (a) avoidance of interpersonal intimacy (α= 0.82), (b) argumentativeness or disagreement (α= 0.74), (c) connection and reciprocity (α= 0.64), (d) conflict aversion (α= 0.72), (e) emotional experience and expression (α= 0.75), and (f) excessive expressivity (α= 0.77). Total score of FIAT-Q-SF had mean -16.56 and a standard deviation (SD) of 18.31 in its validation study. Values 1-SD above the mean are considered worse interpersonal functioning while scores 1-SD below of the mean are considered improvements in social functioning.
Depression Anxiety Stress Scale (DASS-42) | Through study completion, an average of 1 year
  DASS is a 42-items self-report scale developed to measure emotional states of depression, anxiety, and stress over the past week. The sum of DASS-42 scales provides an estimate of psychological distress. DASS has shown a consistent three-factorial structure, as well as convergent and discriminant validity. DASS total score and their sub-scales have found a good reliability using the Cronbach's alpha: depression α=0.947, anxiety α=0.897, stress α=0.933, and total score α=0.96. The following cutt-off points for each category of the DASS based on normative percentiles: (a) normal (0-78 percentile), (b) mild (78-87 percentile), (c) moderate (87-95 percentile), (d) severe (95-98 percentile), and (e) extremely severe (98-100 percentile). Scores above 78 percentile in one or more of DASS sub-scales are indicative of psychological distress.
Changes in clients Behaviors and therapists responses in session | Through study completion, an average of 1 year
  Frequency of clients and therapists' behaviors in session will be assessed coding therapeutic interactions. Functional Analytic Psychotherapy Rating Scale (FAPRS) is a coding system designed for assessing behaviors within the clinical setting based on behavior analytic principles. Trained coders will rate the presence or absence of FAPRS codes on a turn-by-turn basis. This allows researchers to evaluate the mechanisms of change of FAP and therapists' adherence to FAP procedures (providing contingencies of reinforcement).

SECONDARY OUTCOMES:
Working Alliance Inventory-Short Revised (WAI-SF) | Through study completion, an average of 1 year
  WAI-SF is a 12-items self-report inventory developed to characterize the therapeutic relationship. This instrument assesses therapist and client's feelings and attitudes regarding goals (objectives of therapy), tasks (agreement of the tools and strategies used by the therapist to reach the therapeutic goals), and bonds (quality of the relationship between therapist and client). WAI-SF has shown a good fit model for a three-factor structure. The total score and the three subscales have found a good reliability using the Cronbach's alpha: goal α=0.87, task α=0.85, bond α=0.80, and total score α=0.91. Higher scores on the WAI-SF indicate a better therapeutic relationship while lower scores indicated worse therapeutic alliance.
The Functional Analytic Psychotherapy-Intimacy Scale (FAP-IS) | Through study completion, an average of 1 year
  FAP-IS is a 14-item scale developed for assessing intimacy related behaviors based on a behavioral analytic conceptualization. This instrument assesses three main components of intimacy: hidden thoughts and feelings (5 items), expression of positive emotions (4 items), and honesty and genuineness (5 items). FAP-IS factors demonstrated a moderate to strong relation each other and presented good to excellent internal consistency using the Cohen's alpha: hidden thoughts and feelings α=0.86, expression of positive emotions α=0.93, and honesty and genuineness α=0.92. The FAP-IS total also showed an excellent reliability index (α= 0.91). A total score of intimacy is obtained by summing all items scores. Finally, higher scores in this scale indicate a high level of intimacy while lower scores indicate poor intimacy.

CONTACTS AND LOCATIONS:
Overall Officials: William C Follette, Ph.D., Principal Investigator — University of Nevada, Reno
Locations (1):
- University of Nevada, Reno, Reno, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share all IPD that underlie results in a publication such as unidentifiable questionnaires and coding raw data. Data that contain HIPAA protected information (e.g., video records) won't be shared to other researchers.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: It is planned that IPD and additional supporting information will become available by June 2019 for 5-year (June 2024).
Access Criteria: IPD and additional supporting information will be shared for publication and replication purposes. They will be only available in protected databases and for scientific purposes.

REFERENCES:
- [Background] Borckardt JJ, Nash MR. Simulation modelling analysis for small sets of single-subject data collected over time. Neuropsychol Rehabil. 2014;24(3-4):492-506. doi: 10.1080/09602011.2014.895390. Epub 2014 Mar 19. PMID 24641472
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Leonard, R. C., Knott, L. E., Lee, E. B., Singh, S., Smith, A. H., Kanter, J., Norton, P.J., & Wetterneck, C. T. (2014). The development of the functional analytic psychotherapy intimacy scale. The Psychological Record, 64, 647-657. DOI10.1007/s40732-014-0089-9.
- [Background] Callaghan, G. M., Follette, W. C., Ruckstuhl, L. E., Jr., & Linnerooth, P. J. N. (2008). The Functional Analytic Psychotherapy Rating Scale (FAPRS): A behavioral psychotherapy coding system. The Behavior Analyst Today, 9, 98-116. DOI: http://dx.doi.org/10.1037/h0100648
- [Background] Callaghan, G. M. (2006). The Functional Idiographic Assessment Template (FIAT) system: For use with interpersonally-based interventions including Functional Analytic Psychotherapy (FAP) and FAP-enhanced treatments. The Behavior Analyst Today, 7, 357-398. http://dx.doi.org/10.1037/h0100160.
- [Background] Darrow SM, Callaghan GC, Bonow JT, Follette WC. The Functional Idiographic Assessment Template-Questionnaire (FIAT-Q): Initial Psychometric Properties. J Contextual Behav Sci. 2014 Apr 1;3(2):124-135. doi: 10.1016/j.jcbs.2014.02.002. PMID 25250219
- [Background] Hedges LV, Pustejovsky JE, Shadish WR. A standardized mean difference effect size for single case designs. Res Synth Methods. 2012 Sep;3(3):224-39. doi: 10.1002/jrsm.1052. Epub 2012 Aug 14. PMID 26062165
- [Background] Kohlenberg, R. J., & Tsai, M. (1991). Functional Analytic Psychotherapy: A guide for creating intense and curative therapeutic relationships. New York: Plenum.
- [Background] Marso, D., and Shadish, W.R. (2014). User Guide for DHPS, D_Power, and GPHDPwr SPSS Macros (Version 1.0). Unpublished manual available from: http://faculty.ucmerced.edu/wshadish/software/software-meta-analysis-single-case-design.